CLINICAL TRIAL: NCT01115764
Title: LV Diastolic Dysfunction Among the Patients With Systolic Heart Failure
Brief Title: LV Diastolic Dysfunction Among the Patients With Systolic Heart Failure-clinical Significance and Prognostic Importance.
Acronym: dd
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: MeirMc, Israel, : Helsinki Committee, MeirMc, Israel
Other Study IDs: MMC10023/2010kCTIL
Record Dates: First submitted 2010-05-02; First posted 2010-05-04 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Heart Failure
Keywords: diastolic dysfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aims: To test the hypothesis that Diastolic dysfunction severity correlates with adverse clinical outcome in patients with systolic heart failure.

DETAILED DESCRIPTION:
Recent studies have explored the prognostic role of TDI-derived parameters in major cardiac diseases, such as heart failure, acute myocardial infarction, and hypertension.(1-3). In these conditions, myocardial mitral annular or basal segmental (Sm) systolic and early diastolic (Ea or Em) velocities have been shown to predict mortality or cardiovascular events. In particular, those with reduced Sm or Em values of <3 cm/s have a very poor prognosis. In heart failure and after myocardial infarction, noninvasive assessment of LV diastolic pressure by transmitral to mitral annular early diastolic velocity ratio (E/Ea or E/Em) is a strong prognosticator, especially when E/Ea is > or =15. (3) Conventional Doppler indices and TDI parameters correlated with functional class in patients with advanced heart failure. The E/E' ratio, which probably reflects high LV end-diastolic pressure, was the best measure for differentiating patients with functional class III and IV, and it also correlated with cardiac mortality and hospitalization for worsening heart failure, thereby providing additional value to standard echocardiographic measures(4-5) In our study we'll try to demonstrate that clinical deterioration of patients with LV systolic dysfunction directly correlates with parameters of their diastolic function and that these parameters more predictable than changes in LVEF.

This study will be performed on the base of Natania Heart Institute (out of hospital clinic).

Within community-based population study we'll select the patients with LV systolic dysfunction.

The participants will be classified according to their LV systolic function, functional class (NYHA) of HF.

Approximately 200 subjects will be enrolled.

The participants will be evaluate according their baseline features, clinical status using EQ-5D score, KCCQ Overall Summary Score, KCCQ Symptom Frequency Score.

After enrolment all our patients will undergo:

1. Maximal work capacity testing (in METS) per BRUCE protocol,
2. HR response estimation,
3. 6-min walk test (to walk down 100 foot corridor to cover as much as possible in 6min)
4. VO2 estimation using the knowing formula VO2 (mlO2/kg/min) = (mphX2.68)+(1.8X26.82XmphXgrade+100)+3.5 1MET =3.5 ml Q2/kg/min
5. Echocardiography will be performed by VIVID -7 with 3.7 MHz probe All subjects examined with color TDI, FPV, two-dimensional and M-mode echo in the left lateral decubitus position.

Follow-up Follow-up at least 2 years With out patients clinical evaluation monthly Exercise capacity evaluation every 3 mo Echocardiography one in half a year

ELIGIBILITY:
Summary of Subject Eligibility criteria:

* Men and women >18 years of age.
* HF of> 3 mo duration and NYHA class II, III, or IV at time of randomization.
* LVEF <45%
* Blood pressure <160/100
* No HF primarily due to valvular heart disease and no clinically significant valvular heart disease that might lead to surgical correction within 12 months of randomization.
* No implantable ICD or CRT within 30 days prior to randomization.
* No chemo- or radio-therapy for treatment of a malignancy within 6 months prior to randomization or clinical evidence of current malignancy with the following exception: local BCC of the skin or cervical intraepithelial neoplasia.
* Serum creatinine<2.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population
  This study will be performed on the base of Natania Heart Institute (out of hospital clinic).
  Within community-based population study we'll select the patients with LV systolic dysfunction.
  The participants will be classified according to their LV systolic function, functional class (NYHA) of HF.
  Approximately 200 subjects will be enrolled.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
-Time to death from any cause or fist hospital admission for worsening HF, whichever occurs fist. | 2 y
  Follow-up -2 y With out patients clinical evaluation monthly Exercise capacity evaluation every 3 mo Echocardiography one in half a year

SECONDARY OUTCOMES:
Change from baseline to month 6 : in KCCQ Overall Summary Score | 6 mo
  Change from baseline to month 6 :
  in KCCQ Overall Summary Score
  in KCCQ Symptom Frequency Score.
  of EQ-5D
  in NYHA class of each time- point.
  in maximal work capacity
  in 6-min walk test
  Change in VO2
  Total number of hospital admission for worsening HF
  Total duration of hospital admission for worsening HF
  Total number of hospital admission for non-fatal c-v event, resuscitated sudden death, arrhythmia, new onset atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Korotinsky Svetlana, doctor, Principal Investigator — Israel: Clalit Health Services